CLINICAL TRIAL: NCT01542112
Title: An Innovational Model to Manage Patient Expectations and Improve Patient Satisfaction: An Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Patient-Centered care; AUH (Other: Aarhus University Hospital)
Record Dates: First submitted 2012-02-13; First posted 2012-03-02 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Patient-Centered Care; Patient Satisfaction
Keywords: Patient-Centered Care; Patient Satisfaction; Interventional study; Patient Expectations; Hospitalization
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PSactive model (Experimental): The model is designed to address the main issues that lie at the core of initiatives to manage patient expectations and improve patient satisfaction. It is a structured interventional set of activities, which gives the clinician an opportunity to meet patient expectations and improve patient satisfaction.
  The interventional model is comprised of teachable-learnable interpersonal communicative steps occurring between the clinician and the patient which are: Gather information on the patient's expectations and perception of the hospitalization, respond, provide relevant information and document the intervention.
  Interventions: Other: PSactive model
- No treament (Experimental): Usual routine in the department
  Interventions: Other: No treatment

INTERVENTIONS:
Other: PSactive model — The model is designed to address the main issues that lie at the core of initiatives to manage patient expectations and improve patient satisfaction. It is a structured interventional set of activities, which gives the clinician an opportunity to meet patient expectations and improve patient satisfaction.
  The interventional model is comprised of teachable-learnable interpersonal communicative steps occurring between the clinician and the patient which are: Gather information on the patient's expectations and perception of the hospitalization, respond, provide relevant information and document the intervention.
  Arms: PSactive model
Other: No treatment — Patients in this arm receive the usual routine in the department.
  Arms: No treament

SUMMARY:
This new model to manage patient expectations was developed based on our international study conducted in four countries. The model is designed to address the main issues that lie at the core of initiatives to manage patient expectations and improve patient satisfaction. It is a structured interventional set of activities, which gives the clinician an opportunity to meet patient expectations and needs and thereby, improve patient satisfaction.

The interventional model comprise teachable-learnable communicative steps occurring between the clinician and the patient which are: Gather information on the patient's expectations and perception of the hospitalization, Respond, Provide relevant information and Document the intervention.

The intervention includes all frontline care givers; however, most of the activities will be done by the nursing staff. The set of activities will be executed by the nurses at three separate periods of time during the patient's hospitalization: time of admission, intermediate time and at time of discharge.

The study is based on the hypothesis that a structured interventional model will significantly improve patient satisfaction during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* all patient older than 17 years who are able to express their expectations and needs to the clinicians and further have the ability to understand and fill in a questionnaire

Exclusion Criteria:

* Patients who are demented

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 835 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Level of satisfaction with the hospitalization. | A questionnaire will be handed directly to the included patients after discharge has been ordered by a physician. The time frame for outcome measuring is anticipated to be within an average of 1-6 hours before the patient leaves the department.
  We will use the Danish National Patient Satisfaction Survey Instrument(20 questions)supplemented with 17 validated questions related to patient expectations, satisfaction and demographic data.
  The primary question is:
  In general, to what extent did your entire experience during the hospitalization meet your expectations? Using any number from 0 to 10, where 0 represents that your expectations were completely unmet and 10 represents that your expectations were completely met - what number would you use to rate this hospital stay?

CONTACTS AND LOCATIONS:
Overall Officials: Ronen Rozenblum, PhD, Principal Investigator — Division of General Internal Medicine, Brigham and Womens Hospital, Harvard Medical School, 1620 Tremont Street, BS-3, Boston 02120, USA
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Rozenblum R, Lisby M, Hockey PM, Levtizion-Korach O, Salzberg CA, Lipsitz S, Bates DW. Uncovering the blind spot of patient satisfaction: an international survey. BMJ Qual Saf. 2011 Nov;20(11):959-65. doi: 10.1136/bmjqs-2011-000306. Epub 2011 Sep 22. PMID 21949436